CLINICAL TRIAL: NCT03629015
Title: The Safety Study of Stemchymal® (Allogeneic Adipose-Derived Mesenchymal Stem Cells) Treating on Acute Liver Failure - An Open-Label, Single-Center Phase I Trial
Brief Title: Safety Study of Stemchymal® in Acute Liver Failure
Acronym: ALF
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Corporate strategic consideration
Sponsor: Steminent Biotherapeutics Inc. (Industry)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AA01
Record Dates: First submitted 2018-07-30; First posted 2018-08-14 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Stem Cells; Adult Stem Cells; Acute Liver Failure; Acute-On-Chronic Liver Failure; Steminent
MeSH Terms: conditions — Liver Failure, Acute; Acute-On-Chronic Liver Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stemchymal® (Experimental): Biological: Stemchymal® ALF/ ACLF patients will receive low (0.5 x 10^6 cells/kg) or high (2 x 10^6 cells/kg) dose of Stemchymal® through intravenous infusion
  Interventions: Biological: Stemchymal®

INTERVENTIONS:
Biological: Stemchymal® — ALF/ ACLF patients will receive Stemchymal® through intravenous infusion

SUMMARY:
To investigate the safety of Stemchymal® via intravenous (IV) infusion in acute liver failure (ALF) and acute on chronic liver failure (ACLF) patients.

ELIGIBILITY:
Inclusion Criteria:

1. ALF or ACLF patients.
2. Subjects are between 20 and 70 years of age.
3. MELD scores meet 17 ≤ MELD ≤ 26.
4. Subjects who had completed signing informed consent.

Exclusion Criteria:

1. Subjects who had been enrolled in any other cell therapy within six months.
2. Females with a positive pregnancy test result.
3. Subjects have contraindication for liver transplantation.
4. Subjects with psychiatric illnesses.
5. Subjects who are diagnosed as active tuberculosis (TB).
6. Subjects with immunological disorders (e.g. autoimmune hepatitis) or using immunosuppressive drugs (e.g. steroid for immunosuppression) within six months prior to screening visit.
7. Subjects with unstable illnesses or contraindication for this clinical trial according to investigator's judgment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AEs) and suspected unexpected serious adverse reaction (SUSAR) | 12 months

OTHER OUTCOMES:
Changes of Model for End-Stage Liver Disease score | 12 months
Changes of Child-Pugh score | 12 months
Changes of Eastern Cooperative Oncology Group performance scale | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No